CLINICAL TRIAL: NCT00402779
Title: Erlotinib Prevention of Oral Cancer (EPOC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2003-0824; EPOC; P01CA106451 (NIH); NCI-2009-00873 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Oral Cancer
Keywords: Oral Cancer; Oral IEN Lesion with LOH; Loss of Heterozygosity; Intraepithelial Neoplasia; Placebo; Erlotinib; Tarceva; OSI-774
MeSH Terms: conditions — Mouth Neoplasms; Carcinoma in Situ | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erlotinib (Experimental): Balanced randomization: Erlotinib 150 mg continuous administration for 1 year.
  Interventions: Drug: Erlotinib
- Placebo (Placebo Comparator): Balanced randomization: Placebo continuous administration for 1 year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib — 150 mg by mouth daily
  Other Names: Tarceva; OSI-774
  Arms: Erlotinib
Drug: Placebo — Tablet by mouth daily
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if erlotinib hydrochloride (Tarcevaâ (OSI-774 ) can prevent cancer in the mouth of people with a high risk of developing cancer in the mouth. The safety of this drug will also be studied, as well as the drug's effect on different cells in the body.

DETAILED DESCRIPTION:
Erlotinib hydrochloride is designed to block the activity of an enzyme found on the surface of many tumor cells that may control tumor growth and survival. This may keep tumors from growing.

If you are found to be eligible to participate in the study, you will be randomly assigned (as in the toss of a coin) to receive either erlotinib hydrochloride or placebo. A placebo is a substance that looks like the study drug but has no active ingredients. Neither you nor the investigators will know which treatment group you have been assigned to. However, in the event of a medical emergency, the study chair can find out which group you are in, if necessary. You can be informed which of the groups you were assigned to, after the study has ended. There is no certainty that you will have an effect from the treatment, or if you will be placed in a group with the active study drug.

While on study, you will take the study dose (either erlotinib hydrochloride or placebo) by mouth, in tablet form, once a day. Tablets should be taken in the morning 1 hour before or 2 hours after a meal, other medications, vitamins, and iron supplements, with no more than 7 ounces of water. You should take the study dose around the same time every day. Every attempt should be made to keep from vomiting the dose, for at least 30 minutes after taking it. For example, if you feel nauseated before or after taking the study dose, anti-nausea medications should be used. If you vomit after taking the study dose, the dose can be taken again only if the tablet(s) can actually be seen and counted (in other words, they have not dissolved yet). You will need to note the time you take each dose of medication throughout the study on a calendar that the study nurse will give to you.

At Months 1, 3, 6, 9, and 12, you will return to clinic. You will have a physical exam including measurement of vital signs. You will have a careful examination of the inside of your mouth.You will have blood (about 2 teaspoons) drawn for routine tests and to check your liver function (about 1-2 teaspoons). At Months 3, 6, and 12, you will have blood (about 2 teaspoons) drawn for research testing and to measure the level of study drug in the body.

Your study doctor will ask you about any medications you are taking, how you are feeling (symptoms), and your current smoking and alcohol usage.

The nurse or study coordinator will collect the medication you did not take, as well as your completed pill diaries, at every clinic visit. At Months 1, 3, 6, and 9, you will also be given new study medication and pill diaries.

You may also have another small biopsy performed from the inside of your mouth in the area where the cells that might become cancerous are located. The biopsy will be performed by your doctor and will be sent to a lab for testing. At months 3 and 12, the doctor will also count and measure any red or white patches on the inside of your mouth. Biopsies will be taken after 3 months of treatment and at the end of 12 months of treatment. The tissue will be tested to see if there are any cells that might become cancerous.

Following the end of treatment, you will return to the clinic every 6 months for 2 years. You will have a complete physical exam, including measurement of vital signs. You will have a careful examination of the inside of your mouth. You will have blood drawn (about 2 teaspoons) for routine tests, to check your liver function, and for research testing. Your study doctor will ask you about any medications you are taking and how you are feeling (symptoms), and your current tobacco and alcohol use.

In addition, at the final clinic visit, you will also take part in a personal interview. During the interview, you will be asked questions regarding socio-demographic information (such as age and race), nutrition habits, current and earlier tobacco use, alcohol use habits, family history of cancer, use of medications, and how you are feeling. The interview will take about 90 minutes to complete. The purpose of the interview is to collect information to learn if there is a relationship between certain factors and your risk of developing cancer of the mouth. You may be contacted in the future in order to collect more information.

You may be taken off study if you are not able to follow the doctors' instructions, serious side effects occur, or the doctor thinks it is in your best interest to leave the study. If you are taken off study for any reason, you will be asked to return to the clinic for a final clinic visit, preferably within 14 days after leaving the study.

This is an investigational study. Erlotinib hydrochloride is approved by the FDA for treatment of NSCLC. Its use in this study is considered investigational. Approximately 491 patients will be screened for this study. Up to 120 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with one of the following: (a) loss of heterozygosity (LOH) at 3p14 and/or 9p21 in the oral IEN of patients with a history of curatively treated oral cancer or (b) LOH at 3p14 and/or 9p21 plus at one other chromosomal region in the IEN of patients with no oral cancer history.
2. Participants must have confirmed diagnosis of oral IEN lesion with LOH. (Note:The initial screening biopsy of oral IEN lesion with LOH must be obtained within 12 months of study enrollment. If initial diagnostic biopsy for LOH is > 3 months prior to study enrollment, investigators may use clinical judgment to order an additional screening biopsy to assess histopathological changes).
3. Age >/= 18 years
4. ECOG performance status <2
5. Participants must have normal organ & marrow function as defined below w/in 30 days of randomization:CBC w/ differential white cell count-acceptable results must include:WBC >3,000ul, hemoglobin>10 g/dl, platelet count > 125,000ul, LFTs-total bilirubin & alkaline phosphatase, AST (SGOT) & ALT (SPGT) all w/in <1.5xULN.Note:At the discretion of the attending physician,participants w/ Gilbert's disease may still be eligible to participate in the event the total bilirubin value is >1.5xULN. Kidney function-serum creatinine< 1.5xULN Chemistry-Sodium & potassium all w/in normal institutional limits.
6. The effects of the study agent on the developing human fetus are unknown.For this reason,WOCBP & men must agree to use adequate contraception (hormonal or barrier method of birth control;abstinence)prior to study entry& for the duration of active treatment.Neg.serum pregnancy test in WOCBP.Childbearing potential will be defined as women who have had menses w/in the past 12 mths,who have not had tubal ligation or bilateral oophorectomy.Should a woman become pregnant or suspect she is pregnant while participating in this study,she should inform her study physician immediately
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with active cancer or any cancer within the previous two years, excluding oral and non-melanoma skin cancer.
2. Patients with acute intercurrent illness or who have had surgery, radiation therapy, or chemotherapy within the preceding 4 weeks unless they have fully recovered.
3. Patients with a documented history of coagulopathy and/or those taking warfarin or warfarin-derivative anticoagulants
4. Women who are pregnant (confirmed by b-HCG if applicable) or breastfeeding
5. Any medical or psychological condition or any reason that, according to the investigator's judgment, makes the patient unsuitable for participation in the study
6. Patients who have participated in other experimental therapy studies within 3 months of enrollment to this trial
7. Patients with a history of inflammatory bowel disease
8. Patients with a documented history of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2006-11-03 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Univeristy of Texas M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] William WN Jr, Papadimitrakopoulou V, Lee JJ, Mao L, Cohen EE, Lin HY, Gillenwater AM, Martin JW, Lingen MW, Boyle JO, Shin DM, Vigneswaran N, Shinn N, Heymach JV, Wistuba II, Tang X, Kim ES, Saintigny P, Blair EA, Meiller T, Gutkind JS, Myers J, El-Naggar A, Lippman SM. Erlotinib and the Risk of Oral Cancer: The Erlotinib Prevention of Oral Cancer (EPOC) Randomized Clinical Trial. JAMA Oncol. 2016 Feb;2(2):209-16. doi: 10.1001/jamaoncol.2015.4364. PMID 26540028
- [Derived] Scully C. Challenges in predicting which oral mucosal potentially malignant disease will progress to neoplasia. Oral Dis. 2014 Jan;20(1):1-5. doi: 10.1111/odi.12208. PMID 24320967
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen at the following sites exhibiting oral leukoplakia we approached and enrolled if interested. These include MD Anderson Cancer Center, Memorial Sloan-Kettering, Emory University,the University of Chicago, and the University of Maryland.
Pre-assignment Details: Patients with leukoplakia were screened and, once eligibility was confirmed, patients willing to proceed were randomized to erlotinib or placebo in a double-blinded manner.
Groups:
- Erlotinib: Erlotinib 150 mg PO daily x 12 months
- Placebo: Placebo PO daily x 12 months
Period: Overall Study
Arm/Group | Erlotinib | Placebo
Started | 152 | 151
Completed | 75 | 75
Not Completed | 77 | 76
Not completed — Screen Failure | 77 | 76

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 3 | 2 | 5
  31-40 years | 6 | 9 | 15
  41-50 years | 14 | 13 | 27
  51-60 years | 21 | 25 | 46
  61-70 years | 20 | 22 | 42
  71-80 years | 10 | 4 | 14
  81-90 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 43 | 42 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 70 | 70 | 140
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 68 | 67 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 73 | 75 | 148
  Europe | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Oral Cancer-free Survival in Participants Receiving Erlotinib as Compared With the Control Arm or Placebo Group.
Description: Cancer-free survival defined as time from randomization to the development of histologically confirmed oral cancer.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 75 | 75
Participants | 55 | 18

ADVERSE EVENTS:
Time Frame: From drug start through 30 days after drug discontinuation, an average of 3 years
Arm/Group | Erlotinib | Placebo
All-Cause Mortality (participants affected / at risk) | 6/75 | 6/75
Serious Adverse Events (participants affected / at risk) | 10/75 | 4/75
Other Adverse Events (participants affected / at risk) | 68/75 | 32/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=75) | Placebo (N=75)
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Dehydration (Gastrointestinal disorders) | 1 | 0
Speech Impairment (Nervous system disorders) | 1 | 0
Confusion (Nervous system disorders) | 1 | 0
Dizzines (Nervous system disorders) | 1 | 0
Blurred Vision (Nervous system disorders) | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1
Altered Sexual Function (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=75) | Placebo (N=75)
Anemia (Blood and lymphatic system disorders) | 14 | 20
Decreased Leukocytes (Blood and lymphatic system disorders) | 10 | 0
Fatigue (General disorders) | 46 | 21
Fever (General disorders) | 9 | 0
Insomnia (General disorders) | 9 | 0
Weight loss (Gastrointestinal disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 0
Derm Other (Skin and subcutaneous tissue disorders) | 12 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 13
Pruritis (Skin and subcutaneous tissue disorders) | 49 | 15
Rash (Skin and subcutaneous tissue disorders) | 38 | 19
Rash-acneiform (Skin and subcutaneous tissue disorders) | 65 | 12
Diarrhea (Gastrointestinal disorders) | 68 | 18
Distension (Gastrointestinal disorders) | 5 | 0
Dry mouth (Gastrointestinal disorders) | 9 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 0
Flatulance (Gastrointestinal disorders) | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 14 | 6
Mucositis (Gastrointestinal disorders) | 15 | 7
Epistaxis (Gastrointestinal disorders) | 4 | 0
Rectal bleeding (Gastrointestinal disorders) | 4 | 0
Edema/head and neck (General disorders) | 4 | 0
Elevated Alk Phos (Investigations) | 6 | 0
Elevated ALT (Investigations) | 10 | 13
Elevated Creatinine (Investigations) | 9 | 7
Elevated bilirubin (Investigations) | 16 | 18
Elevated AST (Investigations) | 24 | 0
Hyperkalemia (Investigations) | 11 | 1
Hypomagnesemia (Investigations) | 17 | 0
Hyponatremia (Investigations) | 6 | 0
Dizziness (Cardiac disorders) | 9 | 4
Depression (Psychiatric disorders) | 7 | 0
Dry Eye (Eye disorders) | 0 | 6
Pain (Skin and subcutaneous tissue disorders) | 19 | 0
Pain (Gastrointestinal disorders) | 25 | 24
Pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypertension (Cardiac disorders) | 0 | 6
Nausea (Gastrointestinal disorders) | 0 | 12
Sinus Infection (Infections and infestations) | 0 | 4
Headache (General disorders) | 0 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-05-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT00402779/Prot_SAP_000.pdf